CLINICAL TRIAL: NCT06322966
Title: Learning and Living With Wildfire Smoke: Creating Air Clean Environments in Schools Through Youth Participatory Action Research
Brief Title: Learning and Living With Wildfire Smoke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Savannah D'Evelyn, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00017745; K99ES034442 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-03-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Behavior and Behavior Mechanisms; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Air Action Curriculum — The goal of integrating a new curriculum into classrooms is to improve student knowledge on the health effects of air pollution, specifically of wildfire smoke.
  The goal is to implement a student-designed and student-driven air quality study in each school that will lead to improved air quality and health impacts in schools, promote health equity, and train young people to be more informed about their health and proactive citizens in their school community and beyond.
  Other Names: YPAR monitoring project

SUMMARY:
The proposed intervention in this Youth Participatory Action Research (YPAR) proposal will improve knowledge and awareness of the health impacts of air pollution exposure, will elevate the youth voice, improve youth self-efficacy and lead to behavior changes that would reduce exposure to air pollution in a high school setting. These outcomes will be accomplished through the introduction of a new air quality curriculum into science classes, and the establishment of an after-school air quality monitoring program.

All students enrolled in Food Science (Montrose High School), Intro to Agriculture (The STEAD School) and Environmental Science Academy (Grand Junction High School) will participate in the new air quality curriculum, as it will be built into the existing lesson plans. For the after-school monitoring program, the PI and participating teachers (Letters A and B) will recruit 10 to 15 students at each school to be involved in the Student Research Cohort (SRC). Information on this program and how to apply will be shared with students through their health and science classes, included in the school newsletter, and posted on billboards around the school. Students will be identified within the following inclusion criteria: 1) freshman or sophomores in high school and 2) participation in the air quality curriculum. New students will be recruited each year to keep a consistent group as students leave and/or graduate. New students will be brought up to speed by carry-over students, and each new year will represent a separate SRC dedicated to a specific goal.

DETAILED DESCRIPTION:
Air Quality Curriculum: The goal of integrating a new curriculum into classrooms is to improve student knowledge on the health effects of air pollution, specifically of wildfire smoke. The curriculum was jointly designed by the PI and colleagues at CO Dept of Public Health and Environment to teach at the intersection of air pollution, citizen science and civic action and to create critical thinkers who understand they can impact air quality in their community. Students will learn research and air quality 101 (with time devoted specifically to wildfire smoke), learn to measure both their personal exposure to air pollutants and acute health outcomes of exposure, and will be taught the basics of sensors and of air quality monitoring networks. The PI will be available to assist in teaching any lessons as necessary.

YPAR Air Quality Monitoring Project: The goal of the SRC is to implement a student-designed and student-driven air quality monitoring study. Based on the knowledge they gained from the curriculum, and given access to outdoor, indoor, and personal monitoring devices, the SRC will pose research questions, design a study to answer these questions, and collect and analyze data to share with their school community.

Students will begin this portion of the project by developing research questions that will address air quality issues in each school community. The PI will support students in developing questions that would fill research gaps about: a) wildfire smoke versus other pollutant sources; b) indoor-outdoor infiltration; and c) exposure differences throughout the school building and or throughout a student's day. Once 3-5 questions have been developed, students will be given a list of materials (three-five indoor stationary monitors, one-two outdoor stationary monitor and five handheld mobile monitors), information about any constraints (Wi-Fi availability; facilities restrictions) and a manual for monitor setup. The manual will support students in placing monitors, teach them how to calibrate and maintain monitors, how to process data for QA-QC, and how to analyze monitor data. The SRC will then develop a research plan and place monitors in locations that will allow them to answer their research questions. Once the plan is solidified and approved by the PI, students will present their plan to school administrators and facilities staff to ensure feasibility of monitor placement. To encourage self-efficacy and engagement with the systems of power in their school community, the meeting to present their plan will be arranged by the students themselves. In this meeting, students will present the questions they wish to answer, their plan to do so, and ask for any assistance they may need from facilities (power sources) or IT (Wi-Fi access) in order to begin data collection.

Impact of student participation: The impact on students of the curriculum and involvement in the SRC will be separately evaluated to measure both student's content knowledge, self-efficacy and behavior through both qualitative and quantitative data collection.

To measure the impact of the curriculum quantitatively, a Likert-style survey will assess 1) content knowledge based on completion of the curriculum learning objectives, and 2) student self-efficacy using the Sociopolitical Control Scale (SPCS) for Youth. Content knowledge questions will ask students to rank the extent of understanding for each learning objective and the self-efficacy questions will use the established SPCS for youth to measure students' self-perceptions in two domains: 1) capacity to organize a group of people to achieve certain goals; and 2) ability to influence decisions in their community. Both the content knowledge and self-efficacy portions of the Likert-style survey will be given to all students participating in the curriculum before and after the curriculum lessons (beginning and end of semester). Qualitative data will also be collected via a reflective memo on student interactions and learning written at the end of every curriculum lesson by teachers. The PI will create a template for reflective memos to lessen the burden on teachers, and to ensure the memo is specific to both the learning objectives and the SPCS for youth.

A similar approach will be used to measure the impact of participation in the SRC. As all of the students participating in the SRC will have participated in the air quality curriculum, the quantitative assessment for this group will focus solely on self-efficacy and behavior change. The self-efficacy portions of the quantitative, Likert-style survey will be given to all SRC students at the beginning and end of each school year. Additionally, SRC-generated artifacts (notes and journals) will be collected continuously throughout the year for qualitative analysis.

An additional Likert-style survey will be given to all students (SRC and curriculum only students) in the final year of the grant to assess the impact of the curriculum and monitoring program on air-quality related behavior changes overall. The purpose of these surveys will be to evaluate content knowledge on the health effects of smoke exposure, as well as changes in individual and school-wide behaviors post-implementation of the intervention plan. This survey will be Likert-style and a combination of 1) a series of questions developed to assess comprehension of new knowledge specific to the intervention; and 2) validated questions from the 2007-2011 NHANES survey to evaluate behavior change specific to air quality. Questions include the following themes: mask use; time outdoors versus indoors; exercise schedule; transportation and air filtration.

ELIGIBILITY:
Inclusion Criteria:

* Freshman and Sophomore students at Montrose High School in Montrose, Colorado, Grand Junction High School in Grand Junction, Colorado and the STEAD School in Commerce City, Colorado with the ability to participate for more than two years.
* Teachers, Administrators and Staff at aforementioned high schools willing to participate for more than two years.

Exclusion Criteria:

* Junior and Senior Students at the aforementioned schools (unable to participate for more than two years)
* Teachers, Administrators and Staff at aforementioned high schools unwilling or unable to participate for more than two years.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Number of students, staff, teacher and administrators with higher scores on a Likert-style questionnaire for content knowledge learning objectives. | Year 1 and 2
  Improved Health Knowledge, Attitudes and Practice related to the health impacts of local air pollution across students, staff, teachers and administrators are measured pre and post involvement in an air quality curriculum intervention via a likert scale survey to measure predetermined learning objectives.
Scores on Likert-style questionnaire to evaluate behavior change around air quality. | Year 3 and 4
  A Likert-style survey will be given to all students to assess the impact of the curriculum and monitoring program on air-quality related behavior changes post-intervention. (The air quality intervention is to be designed by students as part of the project but could include interventions such as changes to filtration systems, an anti-idling or educational campaign.) The Likert-style survey will be validated questions from the 2007-2011 NHANES survey to evaluate behavior change specific to air quality. Questions include the following themes: mask use; time outdoors versus indoors; exercise schedule; transportation and air filtration.
Change in student exposure to air pollution calculated through measurements of indoor particulate matter and indoor carbon dioxide. | Year 4 and 5
  Indoor air quality levels (particulate matter and carbon dioxide) will be measured with indoor air quality sensors before and after each air quality intervention plan (such as changes to filtration systems, an anti-idling or educational campaign) has been implemented. Overall student exposure is calculated with approximate respiratory rates and time spent in each indoor location.

CONTACTS AND LOCATIONS:
Overall Officials: Savannah D'Evelyn, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided